CLINICAL TRIAL: NCT06339853
Title: A Single-arm Clinical Trial to Evaluate the Safety and Efficacy of Digital Cognitive Behavioral Therapy With Wearable Device for Insomnia
Brief Title: Study of Efficacy of Digital Cognitive Behavioral Therapy With Wearable Device for Insomnia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1-2023-0023
Record Dates: First submitted 2024-03-17; First posted 2024-04-01 (Actual); Last update posted 2024-04-01 (Actual); Status verified 2024-03

CONDITIONS: Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Wearable Electronic Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- WELT-IP (Experimental): Eligible subjects were able to access WELT-IP (an investigational digital therapeutic) on a mobile device (iOS and Android) as scheduled to receive cognitive behavioral therapy for insomnia (CBT-I). To collect sleep and environmental data, participants will wear the wearable devices, either (1) Apple Watch (Apple Watch Series 8 41mm (GPS)) or Galaxy Watch 5 40mm (Model: SM-R900NZAAKOO), and (2) Oura Ring (Model: Heritage), during the WELT-IP treatment period.
  Interventions: Device: WELT-IP with wearable devices (Apple/galaxy watch. Oura ring)

INTERVENTIONS:
Device: WELT-IP with wearable devices (Apple/galaxy watch. Oura ring) — WELT-IP (an investigational digital therapeutic) is an CBT-I based intervention designed to treat insomnia, conducted in 6 sessions. It is a comprehensive program delivering sleep restriction, stimulation control, muscle relaxation, cognitive treatment, and sleep hygiene education. Main features are sleep diary, sleep reports, daily lessons of CBT-I, muscle relaxation techniques, and cognitive intervention through chatbot. By using WELT-IP simultaneously with wearing an Apple Watch/Galaxy Watch and Oura Ring, sleep and environmental data can be collected.

SUMMARY:
The purpose of the study was to examine safety and efficacy of cognitive behavioral therapy (CBT)-based wearable integrated digital therapeutics for insomnia patients

DETAILED DESCRIPTION:
The investigators intend to conduct a single-arm clinical trial. Following voluntary consent during the screening visit, participants will undergo screening procedures. The screening process will proceed step by step, evaluating selection/exclusion criteria through assessments such as the Mini International Neuropsychiatric Interview (MINI), Columbia Suicide Severity Rating Scale (C-SSRS), etc. Participants who meet the selection criteria and do not meet the exclusion criteria will use the DTx app for 8 weeks. Surveys conducted after app installation (Insomnia Severity Index (ISI), Patient Health Questionnaire-9 (PHQ-9), Generalized Anxiety Disorder 7-item Scale (GAD-7), and a sleep environment questionnaire) will serve as the baseline.

During the clinical trial period, sleep diaries and compliance (lesson completion rate) (applicable only to the experimental group) will be collected through the app. Sleep diaries will be used to evaluate sleep metrics such as sleep efficiency (SE), sleep onset latency (SOL), wake after sleep onset (WASO), etc.

For the experimental group, assessments as per the protocol will be conducted at baseline (Visit 1), and safety (adverse events) evaluation and termination of app usage will occur at 9 weeks (Visit 2).

ELIGIBILITY:
Inclusion Criteria:

1. Individuals aged 19 to 65 years old
2. DSM-5 insomnia disorder patient
3. ISI ≥11
4. Capable of using mobile device and application

Exclusion Criteria:

1. currently on non-pharmacological treatment for insomnia (ex. CBT-I, light therapy, oriental therapy for insomnia)
2. sleep disorders diagnosis other than insomnia (ex. Obstructive sleep apnea, sleep behavior problem, restless leg syndrome)
3. progressive and active medical conditions
4. received continuous psychotherapy such as CBT, motivational enhancement therapy, psychotherapy, and psychoanalysis in the past 3 months
5. major psychiatric illness as assessed through MINI
6. suicide risk as assessed through C-SSRS
7. having occupational risk due to sleep restriction
8. shift workers
9. PHQ-9 of 20 or above
10. Individuals who have actually slept less than an average of 5 hours per night over the past month
11. Pregnant women or individuals planning pregnancy during the clinical trial period

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-09-07 (Actual); Primary Completion 2024-02-29 (Actual); Study Completion 2024-02-29 (Actual)

PRIMARY OUTCOMES:
Change from baseline to week 9 (post-treatment) of ISI | 9 weeks
  Change from baseline to week 9 (post-treatment) of ISI. ISI has 7 questions. Total score ranges from 0 to 28, where higher scores indicate more acute symptoms of insomnia.

SECONDARY OUTCOMES:
Secondary Outcome - Changes from baseline to week 9 of SE | 9 weeks
  Change from baseline to week 9 (post-treatment) of SE. Sleep efficiency is calculated as percentage of total sleep time/time in bed.
Changes from baseline to week 9 of SOL. | 9 weeks
  Change from baseline to week 9 (post-treatment) of SOL. Sleep onset latency is evaluated as the time it takes a person to fall asleep after going to bed.
Changes from baseline to week 9 of WASO. | 9 weeks
  Change from baseline to week 9 (post-treatment) of WASO. WASO is calculated as the total number of minutes that a person is awake after initially falling asleep.
Changes from baseline to week 9 of PHQ-9. | 9 weeks
  Change from baseline to week 9 (post-treatment) of PHQ-9. PHQ-9 has nine questions. Total score ranges from 0 to 27, where higher scores indicate more acute symptoms of depression.
Changes from baseline to week 9 of GAD-7. | 9 weeks
  Change from baseline to week 9 (post-treatment) of GAD-7. GAD-7 has seven questions. Total score ranges from 0 to 21, where higher scores indicate more acute symptoms of anxiety.
Changes from baseline to week 9 of compliance. | 9 weeks
  Compliance (completion rate or lessons) Compliance is evaluated as completion rate of lessons.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Psychiatry, Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Moon DU, Lee Y, Lutt A, Lee S, Lee E. Adjunctive smart ring monitoring during digital cognitive behavioral therapy for insomnia. Sci Rep. 2025 Oct 30;15(1):37934. doi: 10.1038/s41598-025-24312-0. PMID 41168443